CLINICAL TRIAL: NCT03414892
Title: A Phase I Placebo-controlled Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Globalagliatin Hydrochloride After Multiple Ascending Doses in Patients With Type 2 Diabetes Mellitus
Brief Title: Multiple Ascending Doses of Globalagliatin Hydrochloride in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yabao Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YB17071
Record Dates: First submitted 2018-01-07; First posted 2018-01-30 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2018-01

CONDITIONS: Hyperglycaemia (Diabetic); Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Glucokinase Activator
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Globalagliatin Hydrochloride (SY-004) (Experimental): If subjects tolerate 20mg of Globalagliatin Hydrochloride (SY-004) for 7 days, dose escalation will occur in the following order of 40mg, 80mg and 120mg at weekly intervals until patients get intolerant or blood glucose controlled well or reach the maximal dose 120mg.
  Interventions: Drug: Globalagliatin Hydrochloride
- Placebo (Placebo Comparator): If subjects tolerate 20mg of Placebo for 7 days, dose escalation will occur in the following order of 40mg, 80mg and 120mg at weekly intervals until patients get intolerant or blood glucose controlled well or reach the maximal dose 120mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Globalagliatin Hydrochloride — once daily, oral
  Other Names: SY-004
  Arms: Globalagliatin Hydrochloride (SY-004)
Drug: Placebo — once daily, oral
  Arms: Placebo

SUMMARY:
This is a phase I placebo-controlled study to assess safety, tolerability, pharmacokinetics and pharmacodynamics of Globalagliatin Hydrochloride (SY-004) after Multiple Ascending Doses in patients with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
Glucokinase is a characteristic hexokinase isoenzyme in hepatocytes that catalyzes the first step in glucose metabolism. In addition to its role in glucose metabolism, glucokinase is expressed in pancreatic islet beta cells where it acts as a "glucose sensor" for insulin release. Activation of glucokinase increases the glucose sensitivity of insulin secretion, effectively lowering the glucose threshold for insulin secretion. Because of its potential to enhance insulin secretion and affect hepatic glucose metabolism, is being investigated for use as a treatment for hyperglycaemia, Globalagliatin( the active ingredient in SY-004 capsule) is being investigated for use as a treatment for T2DM patients. This is a phase I placebo-controlled study to assess safety, tolerability, pharmacokinetics and pharmacodynamics of Globalagliatin Hydrochloride (SY-004) after Multiple Ascending Doses in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Sex：Male and Female；
2. Age：≥18，≤70；
3. Have T2DM prior to entering the trial based on the disease diagnostic criteria (WHO, 1999), and currently being treated with diet and exercise only or in combined with a stable dose of metformin for at least 8 weeks.
4. 18 kg/m2≤BMI≤35 kg/m2 at screening.
5. 7% ≤ HbA1c ≤11% at screening.
6. 7 mmol/L≤FPG≤13.3mmol/L at baseline.
7. The venous access is normal, and blood samples can be collected according to the protocol.
8. Have given written informed consent to participate in this study.
9. Are well motivated, capable, and willing to communicate with the investigator and complete all the requirements according to the protocol.

Exclusion Criteria:

1. Personnel and their direct relatives of the clinical research unit and its related facilities. Direct relatives mean all biologically and by law related relatives, including spouse, parent, child and sibling,
2. Have been diagnosed with type 1 diabetes, or gestational diabetes mellitus, or a specific type of diabetes mellitus.
3. Clinically significant coronary events or symptoms within 6 months prior to study entry.
4. Clinically significant peripheral vascular disease.
5. Clinical evidence of active diabetic proliferative retinopathy.
6. Known clinically significant autonomic neuropathy as evidenced by urinary retention, orthostatic hypotension, diabetic diarrhea or gastroparesis.
7. With a history of diabetes or diabetic ketoacidosis, lactic acidosis, hyperosmolar nonketotic coma history.
8. Have severe hypoglycemia occurred before the screening with unknown causes (need other people to help restore) or the frequency of hypoglycemia, such as 3 or more hypoglycemic events(blood glucose ≤3.9mmol/L) within 1 months before screening or hypoglycemia related symptoms.
9. Continuous use of insulin for more than 1 month in last year.
10. Have any disorder or unstable situation of the endocrine system, immune system or other diseases impaired blood sugar(such as Hyperthyroidism, acromegaly, Cushing syndrome) that are required treatment
11. Have significant history of past or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (other than diabetes), hematological, or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs or of constituting a risk when taking the study drug formulations or interfering with the interpretation of data.
12. Have any types of malignancies (whether cured or not).
13. History of haemoglobin disease（such as sickle cell anemia or thalassemia, iron deficiency anemia）.
14. Have known allergies to Globalagliatin or related compounds, or have allergic history, or have taken glucokinase activator in last year.
15. Are currently enrolled in, or discontinued within the last 3 months from, a clinical trial involving an investigational drug or device or use of a drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
16. Have a history of drug or alcohol abuse.
17. Have history of blood donation in last 6 months.
18. Patients who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) (1 unit = 360 mL of beer; 150 mL of wine; 45 mL of distilled spirits) or patients unwilling to stop alcohol consumption 24 hours prior to admission until the completion of each in-patient study period.
19. Patients who smoke >10 cigarettes or other tobacco products per day before study entry. Patients are unlikely / unable to stop nicotine intake during the study period.
20. Fasting serum C peptide< 1.0 ng/ml（333pmol/L）at screening.
21. Patients are treated with stable dose of anti-hypertension drug at least for 4 weeks with inadequate blood pressure control (sitting systolic blood pressure≥160mmHg or diastolic blood pressure≥100mmHg)at screening.
22. QTcB≥450msec at screening.
23. Fasting serum triglycerides>500mg/dL（5.70mmol/L）at screening.
24. ALT (alanine aminotransferase) >1.5 ULN, AST (aspartate transaminase) >1.5×ULN or TBIL (total bilirubin) > 1.5×ULN (UIN :times the upper limit of the reference range)at screening; or have active liver diseases at screening.
25. Serum creatinine>133μmol /L at screening.
26. Use of any known inducers or inhibitors of CYP3A (Cytochrome P450 3A) within 14 days prior to the first dosing with study drug or intended use during the study. Examples of inducers include, but are not limited to, phenytoin, barbiturates, carbamazepine, St. John's Wort, rifampin. Examples of inhibitors include, but are not limited to, fluvoxamine, sertraline, norfloxacin, macrolide antibiotics (erythromycin, clarithromycin), antifungals, human immunodeficiency virus (HIV) protease inhibitors, cyclosporine, diltiazem, pomelo, grapefruit juice.
27. Have been previously enrolled in or withdrawn from this clinical trial.
28. Evidence of positive HBsAg, or IgM (immunoglobulin M ) anti-HBc (hepatitis B core antigen), or anti-HCV (hepatitis C virus ), or anti-HIV, or anti-TPat (treponema pallidum antibody) screening.
29. fertility qualified subjects（Male and Female）are unlikely to use reliable contraception during study period and at least 1 month after last dosing or women in child-bearing age have positive for blood pregnancy tests within 24 hours before enrollment, or pregnant or lactating women.
30. Patients, in opinion of investigator or sponsor, are not suitable for this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
the mean change in glucose area under curve (AUC) from baseline. | 28 days
  Compared with placebo, the mean change in glucose AUC from baseline at D28.

SECONDARY OUTCOMES:
the fasting plasma glucose from baseline | 7, 14, 21, 28 days
  Compared with placebo, the fasting plasma glucose from baseline at D7，D14，D21 and D28.
the changes of MMTT (mixed-meal tolerance test) results from baseline | 28 days
  Compared with placebo, the changes of MMTT (mixed-meal tolerance test) results from baseline at D28
the mean changes of average 7-points blood glucose profiles from baseline | 7, 14, 21, 28 days
  Compared with placebo, the mean changes of average 7-points blood glucose profiles from baseline at D7，D14，D21 and D28.
the mean changes of average 14-points blood glucose profiles from baseline | 7, 14, 21, 28 days
  Compared with placebo, the mean changes of average 14-points blood glucose profiles from baseline at D7，D14，D21 and D28.
the mean changes of post-prandial blood glucose from baseline | 7, 14, 21, 28 days
  Compared with placebo, the mean changes of post-prandial blood glucose from baseline at D7，D14，D21 and D28.

OTHER OUTCOMES:
genetic: TCF7L2 ( Transcription factor 7-like 2) rs7903146 and GCKR (glucokinase regulatory protein) rs780094 ) | 28 days
  The genetic（TCF7L2 rs7903146 and GCKR rs780094）effects on response of SY-004 in T2DM patients.
the changes of GA (Glycated albumin) from baseline | 28 days
  Compared with placebo, the changes of GA (Glycated albumin) from baseline at D28.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Yang, Study Director — Yabao pharmaceutical Group Co.
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng S, Shao F, Ding Y, Fu Z, Fu Q, Ding S, Xie L, Chen J, Zhou S, Zhang H, Zhou H, Chen Y, Sun C, Zhu J, Zheng X, Yang T. Safety, Pharmacokinetics, and Pharmacodynamics of Globalagliatin, a Glucokinase Activator, in Chinese Patients with Type 2 Diabetes Mellitus: A Randomized, Phase Ib, 28-day Ascending Dose Study. Clin Drug Investig. 2020 Dec;40(12):1155-1166. doi: 10.1007/s40261-020-00971-x. Epub 2020 Oct 30. PMID 33125674